CLINICAL TRIAL: NCT05910658
Title: First CRUSH: Piloting the Preliminary Feasibility and Acceptability of the Competence in Romance and Understanding Sexual Health (CRUSH) Curriculum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Susan Faja, Associate Professor, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FP01030935
Record Dates: First submitted 2023-06-01; First posted 2023-06-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-08

CONDITIONS: Autism; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Mental Competency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Other): Participants will receive the CRUSH Curriculum
  Interventions: Behavioral: Competence in Romance and Understanding Sexual Health (CRUSH)

INTERVENTIONS:
Behavioral: Competence in Romance and Understanding Sexual Health (CRUSH) — Manualized curriculum targeting sexual health and behavior in intimate relationships designed to meet the specific needs of autistic adults

SUMMARY:
The goal of this clinical trial is to learn about the feasibility and acceptability of a behavioral intervention in designed to provide sexual education and improve the behavioral skills of autistic adults for intimate relationships.

The main questions it aims to answer are:

* Acquire feasibility and acceptability data for delivery of the CRUSH curriculum in a group didactic setting plus 1-1 coaching.
* Acquire feasibility and acceptability data regarding the assessment battery for future clinical trials.

Participants will complete:

* A screening call.
* Provide documentation of a diagnosis of autism spectrum disorder.
* 3 visits to assess knowledge and behaviors related to dating and sexual health at each point throughout the training curriculum (before beginning, midway, and after finishing).
* 15-20 training sessions to participate in the CRUSH curriculum. After each session, provide feedback about the session.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the feasibility and acceptability of a behavioral intervention in designed to provide sexual education and improve the behavioral skills of autistic adults for intimate relationships, called CRUSH.

The main questions it aims to answer are:

* Acquire feasibility and acceptability data for delivery of the CRUSH curriculum in a group didactic setting plus 1-1 coaching.
* Acquire feasibility and acceptability data regarding the assessment battery for future clinical trials.

Participants will complete:

* A screening call.
* Provide documentation of a diagnosis of autism spectrum disorder.
* 3 visits to assess knowledge and behaviors related to dating and sexual health at each point throughout the training curriculum (before beginning, midway, and after finishing).
* 15-20 training sessions to participate in the CRUSH curriculum. After each session, provide feedback about the session.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 30 years old;
* Documentation of a prior diagnosis of autism spectrum disorder (ASD) or receipt of services based on an ASD diagnosis;
* Ability to provide consent for the protocol and understand task demands (i.e., approximately WASI-2 full scale IQ of 70 or above);
* Fluent in English

Exclusion Criteria:

* Non-English-speaking participants (less than 50% of speech in English);
* Known genetic etiology of ASD (e.g., Fragile X);
* Major mental illness (e.g., bipolar disorder, schizophrenia, or psychosis).
* Live more than 35 miles from Two Brookline Place, Brookline, MA where intervention sessions will be offered.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-10-18 (Estimated)

PRIMARY OUTCOMES:
Acceptability Rating Scale | At baseline enrollment visit and weekly throughout training for a total of 20 weeks
  A measure of the acceptability of methods used in the project including qualitative interview and 5-point rating scale (lower scores indicate higher acceptability)

SECONDARY OUTCOMES:
Feasibility Assessment | At baseline enrollment visit and weekly throughout training for a total of 20 weeks
  Analysis of missing items or session content that cannot be completed (fewer missing items indicates better feasibility)

OTHER OUTCOMES:
Sexual Vocabulary Test | At baseline enrollment visit; 8-10 weeks after beginning intervention (i.e., midpoint); 18-22 weeks after beginning intervention (i.e., post-testing)
  A measure of the ability to provide definitions of sexual health terms to be used as a measure of target engagement (higher score indicates higher level of knowledge)
Mathtech Behavioral Scale | At baseline enrollment visit; 8-10 weeks after beginning intervention (i.e., midpoint); 18-22 weeks after beginning intervention (i.e., post-testing)
  A measure of sexual health and intimate behavior to be used as a primary outcome in a future trial (higher scores indicate higher levels of behavior)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Two Brookline Place, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No